CLINICAL TRIAL: NCT03372408
Title: Parkdale Infant Nutrition Security Targeted Evaluation Project (PINSTEP): Formative Research (Objective 1-Retrospective Chart Review)
Brief Title: Parkdale Infant Nutrition Security Targeted Evaluation Project: Chart Review
Acronym: PINSTEP-1
Status: Completed | Type: Observational
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Sellen, Professor, University of Toronto
Other Study IDs: 34482-1
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Prenatal Community Program; Vulnerable Population; Postnatal Community Program

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Program Clients: Parkdale Parents' Primary Prevention Project (5P's) clients
  Interventions: Other: Chart review

INTERVENTIONS:
Other: Chart review — Retrospective chart review of program participation and socio-demographic & psychosocial characteristics

SUMMARY:
In Toronto Ontario, the Parkdale Community Health Centre operates a community outreach program entitled Parkdale Parents' Primary Prevention Project (5P's). The 5P's provides weekly pre- and post-natal support and education programs for clients. This includes an infant feeding program for mothers with infants 0-6 months (Feeding Tiny Souls). The 5P's has a diverse client-base; the program is aimed at women who are in challenging life circumstances, therefore, clients may include low-income or single mothers and newcomers to Canada.

It is important to know who is accessing community programs and what the drivers of program utilization are in order to better support the women who are enrolled and to target those who are not. The aim of this project is twofold: 1) to investigate what socio-demographic and psychosocial characteristics predict level of participation in a prenatal community outreach program targeting vulnerable mothers and 2) based on utilization of a prenatal program, are there differences in the use of a postnatal program? This study will be conducted through a retrospective chart review. The study population will consist of women who enrolled in 5P's prenatally. The hypothesis is that more vulnerable women will not attend programming as frequently.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Parkdale Parents' Primary Prevention Project (5P's) prenatally
* 5P's client signed the permission to release information on the 5P's intake form

Exclusion Criteria:

* Only attended Parkdale Parents' Primary Prevention Project (5P's) postnatally
* 5P's client did not sign the permission to release information on the 5P's intake form

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Clients enrolled in Parkdale Parents' Primary Prevention Project (5P's) in Toronto, Ontario, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Level of program participation as assessed by review of client records and program attendance records | Registration to prenatal program until 12 months postpartum
  Retrospective chart review of client program records and attendance

CONTACTS AND LOCATIONS:
Overall Officials: Jane Francis, MSc, Principal Investigator — University of Toronto
Locations (1):
- Parkdale Community Health Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] Francis J, Ismail S, Mildon A, Stewart S, Underhill B, Tarasuk V, Di Ruggiero E, Kiss A, Sellen DW, O'Connor DL. Characteristics of vulnerable women and their association with participation in a Canada Prenatal Nutrition Program site in Toronto, Canada. Health Promot Chronic Dis Prev Can. 2021 Dec;41(12):413-422. doi: 10.24095/hpcdp.41.12.02. PMID 34910898